CLINICAL TRIAL: NCT04048317
Title: Effectiveness of Drug Eluting & Conventional Trans-arterial Chemo-embolization in Treatment of Primary Hepatic Cell Carcinoma
Brief Title: Effectiveness of Drug Eluting TACE in Primary HCC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Hassan Taha Abdurabou, Resident radiologist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: effectiveness of TACE
Record Dates: First submitted 2019-07-26; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Hepatic Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin; Ethiodized Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drug eluting bead trans arterial chemo embolization (Experimental): the international arm is the patients embolized with drug eluting bead trans arterial chemo embolization using Hepasphere
  Interventions: Drug: HepaSphere Microspheres/Doxorubicin Hydrochloride
- conventional trans arterial chemo embolization (Placebo Comparator): the control arm is the patients embolized with drug eluting bead trans arterial chemo embolization using Lipiodol
  Interventions: Drug: Lipiodol

INTERVENTIONS:
Drug: HepaSphere Microspheres/Doxorubicin Hydrochloride — evaluation the tumor (size, location and pattern of enhancement) ;and ensure portal vein patency; then evaluation of hepatic arterial anatomy, after that we determine the tumor arterial feeders and the arteries that should be avoided during the maneuver.
  Selective celiac and superior mesenteric angiograms were performed using 5 Fr. Catheter then superselective angiogram were used microcatheter. then injection of drug-eluting microsphere (25 mg Hepasphere 50-100 micron) loaded with 50 mg doxorubicin solution for 2 hours.
  Arms: drug eluting bead trans arterial chemo embolization
Drug: Lipiodol — evaluation the tumor (size, location and pattern of enhancement) ;and ensure portal vein patency; then evaluation of hepatic arterial anatomy, after that we determine the tumor arterial feeders and the arteries that should be avoided during the maneuver.
  Selective celiac and superior mesenteric angiograms were performed using 5 Fr. Catheter then superselective angiogram were used microcatheter. then injection of prepared mixture of Lipiodol and (Doxorubicin or 5-FU) vary in dosage depend on operator consideration
  Arms: conventional trans arterial chemo embolization

SUMMARY:
the aim of this work to compare effectiveness of drug-eluting bead trans-arterial chemo-embolization and conventional trans-arterial chemo-embolization of hepatic cell carcinoma in the aspect of (Tumor response via m-RECIST criteria), (liver injury via Liver function tests and tumor markers) and (survival outcome) of patients treated in Assiut university .

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common cancer in the world and the third most common cause of cancer-related death .. With improved surveillance of patients with chronic liver disease and advances in imaging, more patients are diagnosed with early-stage HCC . For the treatment of early stage HCC, curative therapies including liver transplantation, hepatic resection, and radio frequency ablation (RFA) are recommended. Liver transplantation is the treatment option especially for patients with decompensated cirrhosis, but potential recipients outnumber donors. Hepatic resection is widely used as the main choice of treatment for resectable HCC. However, the risk of postoperative hepatic dysfunction often precludes surgery.

For unresectable patient, trans-arterial chemo-embolization (TACE) was the treatment of choice .

At 2014, Yang et al. compared the treatment effects of hepatic resection, RFA, and conventional TACE on long-term survival. It was found that the range of patients treated by TACE in clinical practice reported survivals widely range from 8-26% at 5-years. which was similar to that with hepatic resection and RFA in patients with single-nodule HCC of 3 cm or smaller without vascular invasion when the underlying liver status was balanced among the patients receiving each treatment. In addition, most of the patients initially treated with c-TACE achieved a complete response, which was one of the independent prognostic factors of survival, although some should receive repeated treatments. However, when c-TACE is used as an initial treatment, special care should be taken to obtain a complete response, and surveillance for tumor recurrence should be undertaken. These results are consistent with those of cohort studies demonstrating that TACE provided overall survival similar to hepatic resection in early-stage HCC .

Conventional (Lipiodol) TACE Base on technique with emulsified combination of chemotherapy such as Doxorubicin and Lipiodol administrate via arterial feeder.

Less in systemic chemotherapy and increase overall survival rate were the most concern in treatment but many studies reported side effects from conventional (Lipiodol) TACE significantly among an improvement of overall survival rate .

Conventional TACE may cause side effects because it can damage healthy cells as it kills cancer cells. Side effects can develop any time during, immediately after or a few days or weeks after chemotherapy . in addition to the patient needed frequent ablation after a short time .

The most commonly Side Effect of TACE is (Post embolization syndrome) which is a group of symptoms . include : fever, Right upper quadrant pain, nausea, vomiting and fatigue .

Other side effects may occur include bruising or bleeding at the catheter site, hair loss, abnormal liver functions, lung infections, gall bladder inflammation and tumor lysis syndrome .

Drug-eluting bead TACE is the new method of delivering chemotherapy during TACE which uses special beads that already have the chemotherapy drug in them . after these are injected into the arteries of the liver , they slowly sustained releasing the drug to treat the tumor .

The studies showed that TACE with (Hepasphere) less systemic side effect in patient than TACE with (Lipiodol) but no definite statistical difference in treatment and survival outcome.

This study compares effectiveness of those methods in treatment of Hepatocellular carcinoma in Assiut university

ELIGIBILITY:
Inclusion Criteria:

* patients must be 18 to 75 years old.
* patients must be diagnosed as primary Hepatocellular carcinoma (HCC) by radiologic imaging revealed angiogenicity pattern .
* All of the patient have Child-Pugh status A or B .
* All of the patient have BCLC stage A or B.
* patients must have adequate renal and liver function accepting the maneuver.
* patients must have adequate coagulation profile (platelets count ≥ 80 000), (prothrombin concentration ≥ 70 %).
* patients must haven't previous history of resection of other ablation (alcohol, radio frequency or micro wave ablation).

Exclusion Criteria:

* patients have previous history of resection of other ablation (alcohol, radio frequency or micro wave ablation).
* patients with impaired coagulation profile (platelets count < 80 000), (prothrombin concentration < 70 %).
* patients with decompensated liver cell failure having ascites which impedes the maneuver .
* patients with past history of reaction to the drug used in maneuver
* patients with poor image quality.
* patients with lost follow up .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of drug-eluting bead trans-arterial chemo-embolization in patients of hepatocellular carcinoma | baseline
  Evaluate the efficacy and safety of drug-eluting bead trans-arterial chemo-embolization in management of HCC patients in comparison of conventional chemo-embolization in 75 stable patients by evaluating the response of embolized lesions for each drug with modified RECIST criteria.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Kudo M, Izumi N, Kokudo N, Matsui O, Sakamoto M, Nakashima O, Kojiro M, Makuuchi M; HCC Expert Panel of Japan Society of Hepatology. Management of hepatocellular carcinoma in Japan: Consensus-Based Clinical Practice Guidelines proposed by the Japan Society of Hepatology (JSH) 2010 updated version. Dig Dis. 2011;29(3):339-64. doi: 10.1159/000327577. Epub 2011 Aug 9. PMID 21829027
- [Background] Zhang BH, Yang BH, Tang ZY. Randomized controlled trial of screening for hepatocellular carcinoma. J Cancer Res Clin Oncol. 2004 Jul;130(7):417-22. doi: 10.1007/s00432-004-0552-0. PMID 15042359
- [Background] Yang HJ, Lee JH, Lee DH, Yu SJ, Kim YJ, Yoon JH, Kim HC, Lee JM, Chung JW, Yi NJ, Lee KW, Suh KS, Lee HS. Small single-nodule hepatocellular carcinoma: comparison of transarterial chemoembolization, radiofrequency ablation, and hepatic resection by using inverse probability weighting. Radiology. 2014 Jun;271(3):909-18. doi: 10.1148/radiol.13131760. Epub 2014 Feb 8. PMID 24520944
- [Background] Salem R, Lewandowski RJ. Chemoembolization and radioembolization for hepatocellular carcinoma. Clin Gastroenterol Hepatol. 2013 Jun;11(6):604-11; quiz e43-4. doi: 10.1016/j.cgh.2012.12.039. Epub 2013 Jan 26. PMID 23357493
- [Background] Hsu CY, Huang YH, Chiou YY, Su CW, Lin HC, Lee RC, Chiang JH, Huo TI, Lee FY, Lee SD. Comparison of radiofrequency ablation and transarterial chemoembolization for hepatocellular carcinoma within the Milan criteria: a propensity score analysis. Liver Transpl. 2011 May;17(5):556-66. doi: 10.1002/lt.22273. PMID 21506244
- [Background] Guo Z, Zhong Y, Hu B, Jiang JH, Li LQ, Xiang BD. Hepatic resection or transarterial chemoembolization for hepatocellular carcinoma within Milan criteria: A propensity score matching analysis. Medicine (Baltimore). 2017 Dec;96(51):e8933. doi: 10.1097/MD.0000000000008933. PMID 29390426
- [Background] Dhanasekaran R, Kooby DA, Staley CA, Kauh JS, Khanna V, Kim HS. Prognostic factors for survival in patients with unresectable hepatocellular carcinoma undergoing chemoembolization with doxorubicin drug-eluting beads: a preliminary study. HPB (Oxford). 2010 Apr;12(3):174-80. doi: 10.1111/j.1477-2574.2009.00138.x. PMID 20590884
- [Background] Lammer J, Malagari K, Vogl T, Pilleul F, Denys A, Watkinson A, Pitton M, Sergent G, Pfammatter T, Terraz S, Benhamou Y, Avajon Y, Gruenberger T, Pomoni M, Langenberger H, Schuchmann M, Dumortier J, Mueller C, Chevallier P, Lencioni R; PRECISION V Investigators. Prospective randomized study of doxorubicin-eluting-bead embolization in the treatment of hepatocellular carcinoma: results of the PRECISION V study. Cardiovasc Intervent Radiol. 2010 Feb;33(1):41-52. doi: 10.1007/s00270-009-9711-7. Epub 2009 Nov 12. PMID 19908093
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- See also: Hepatic Arterial Infusion of Doxorubicin-Loaded Microsphere for Treatment of Hepatocellular Cancer: A Multi-Institutional Registry — https://www.journalacs.org/article/S1072-7515(11)00896-9/abstract